CLINICAL TRIAL: NCT01167426
Title: An Open-Label, Multicenter Study Evaluating Patient Injection Satisfaction With Two Formulations of Glatiramer Acetate (GA) Using Autoject 2 as the Subcutaneous Injection Delivery Method.
Brief Title: Evaluation of Two Glatiramer Acetate (GA) Formulations in Relapsing-Remitting Multiple Sclerosis (RRMS) Patients
Acronym: ENCORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: PM034
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2012-08

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Remitting Multiple Sclerosis; RRMS; Clinically Isolated Syndrome; CIS; Copaxone; glatiramer acetate; Autoject 2
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 20 mg/0.5 mL Glatiramer Acetate (Active Comparator): Participants received once daily subcutaneous administration of 20 mg glatiramer acetate as 20 mg/1.0 mL utilizing autoject 2 for glass syringe for two weeks (Period 1), followed by 20 mg/0.5 mL utilizing the autoject 2 device for four weeks (Period 2).
  Interventions: Drug: Glatiramer Acetate 20 mg/0.5 mL

INTERVENTIONS:
Drug: Glatiramer Acetate 20 mg/0.5 mL — 20 mg/1.0 mL formulation of glatiramer acetate utilizing the autoject 2 for glass syringe.
  Other Names: Copaxone®
Drug: Glatiramer acetate 20 mg/0.5 mL — 20 mg/0.5 mL formulation of glatiramer acetate utilizing the autoject 2 20 mg/0.5 mL device.

SUMMARY:
This is an open-label, multicenter study conducted at approximately 20 sites. Each patient will inject GA daily for 6 weeks utilizing an autoject 2 device to determine overall injection satisfaction.

DETAILED DESCRIPTION:
The study will consist of a 2 week treatment period with participants injecting their current therapy of Copaxone 20 mg/1.0 mL glatiramer acetate utilizing an autoject 2. All participants will then roll over to the new formulation of 20 mg/0.5 mL glatiramer acetate with an autoject 2 device for a 4 week treatment period. Patient satisfaction will be evaluated using an Experience Questionnaire throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with a diagnosis of Relapse Remitting Multiple Sclerosis (RRMS) or Clinically Isolated Syndrome (CIS)
* Currently injecting glatiramer acetate 20 mg/1.0 mL per day subcutaneously (SC) for a minimum of 90 days utilizing the autoject 2 for glass syringe for a minimum of 75% of daily injections
* Willing and able to complete all procedures and evaluations related to the study
* Willing to continue to follow usual injection site preparation and routine adjunctive local injection site reactions (LISR) management techniques
* Willing and able to provide written informed consent

Exclusion Criteria:

* Currently using or treated with another immunomodulating therapy (IMT) in conjunction with GA in the 30 days prior to screening for this study
* Currently using an investigational drug or using treatment with any other investigational agent in the 30 days prior to screening for this study
* Pregnant or planning pregnancy or breastfeeding
* Use of any other parenteral medications (e.g., intramuscular, SC, intravenous, etc.) either currently or in the past 30 days prior to screening for this study
* Any other medical or psychiatric conditions that would make the patient unsuitable for this research, as determined by the Investigator
* Unwilling to perform all daily injections with an autoject 2 device
* Previous participation in any study evaluating the new 20 mg/0.5 mL formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Smith, MD, Study Director — Teva Neuroscience, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Glatiramer Acetate: Participants received once daily subcutaneous administration of 20 mg glatiramer acetate as 20 mg/1.0 mL utilizing autoject 2 for glass syringe for two weeks (Period 1), followed by 20 mg/0.5 mL utilizing the autoject 2 device for four weeks (Period 2).
Period: Overall Study
Arm/Group | Glatiramer Acetate
Started | 148
Completed | 138
Not Completed | 10
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — Sponsor Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Glatiramer Acetate
Number analyzed (Participants) | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 140
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 48.1 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 144
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 141
  Black or African American | 3
  Other | 4
Region of Enrollment [Number; unit: participants]
  United States | 148
Duration of Glatiramer Acetate [Mean (Standard Deviation); unit: years] | 4.823 (3.5539)
Duration of Multiple Sclerosis Disease [Mean (Standard Deviation); unit: years] | 10.167 (9.0643)

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 2 to Week 6 in Composite Score of Patient Satisfaction With Injection Experience
Description: The Satisfaction with Injection Experience questionnaire consists of 5 questions where participants are asked to rate their injection experience over the past 2 weeks on ease of use, bother, acceptability, confidence to inject and satisfaction. The response options range from "strongly disagree" (score = 1) to "strongly agree" (score = 5). The composite score of Satisfaction with Injection Experience is defined as the mean of the five Likert questions. The composite score ranges from 1.0 to 5.0, with a score of 5.0 representing the most satisfaction with injection experience and a score of 1.0 representing the least satisfaction with injection experience.
Time Frame: Week 2 (prior to first injection with 20 mg/0.5 mL formulation), Week 6 (after 4 weeks of treatment with 20 mg/0.5 mL formulation).
Population: The Analysis Population consisted of of all patients who received at least one dose of study medication and had satisfaction data at time points 2 and 6 weeks, 2 and 4 weeks, or 2, 4 and 6 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Glatiramer Acetate
Number analyzed (Participants) | 139
units on a scale
  Week 2 | 4.1 (0.77)
  Week 6 | 4.8 (0.46)
  Change from Week 2 to Week 6 | 0.7 (0.79)
Statistical Analysis 1: Comparison: Glatiramer Acetate; Comparison of Week 2 (20 mg/1.0 mL utilizing autoject 2 for glass syringe) to Week 6 (20 mg/0.5 mL utilizing the autoject 2 20 mg/0.5 mL); Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed-Rank; Difference in mean ranks = 79.6 — Difference in mean ranks between Week 2 and Week 6

2. Secondary Outcome: Patient Injection Experience Preference
Description: The Injection Experience Preference Questionnaire utilizes a 5-level preference scale where participants were asked to compare their injection experience during the first 2 weeks (glatiramer acetate 20 mg/1 mL) with the past 2 weeks (glatiramer acetate 20 mg/0.5 mL). Response options were: 1. "strongly prefer first experience (first 2 weeks)"; 2. "somewhat prefer first experience (first 2 weeks)"; 3. "no preference"; 4. "somewhat prefer second experience (past 2 weeks)"; 5. "strongly prefer second experience (past 2 weeks)." Responses 1 and 2 were combined into a single category (prefers first experience) and responses 4 and 5 were combined into a single category (prefers second experience).
Time Frame: Week 4
Population: Analysis Population with available data.
Measure: Number; unit: participants
Arm/Group | Glatiramer Acetate
Number analyzed (Participants) | 140
participants
  Prefers First Experience | 9 (6.2)
  No Preference | 22
  Prefers Second Experience | 109
Statistical Analysis 1: Comparison: Glatiramer Acetate; Test type: Superiority or Other; p < 0.0001, Chi-squared — Goodness-of-fit p-value comparing overall preference to expected frequencies of 33.3% in each category. That is, no preference across the full sample of patients in the study

ADVERSE EVENTS:
Description: All patients who receive at least 1 dose of study medication were included in the Safety population. 148 patients were exposed to the 20 mg/1.0 mL formulation of glatiramer acetate utilizing the autoject 2 for glass syringe and 142 patients were exposed to the 20 mg/0.5 mL formulation utilizing the autoject 2 20 mg/0.5 mL device.
Groups:
- Period 1: Glatiramer Acetate 20 mg/1.0 mL: Participants received once daily subcutaneous administration of 20 mg glatiramer acetate as 20 mg/1.0 mL utilizing autoject 2 for glass syringe for two weeks (Period 1).
- Period 2: Glatirimer Actetate: Participants received once daily subcutaneous administration of glatiramer acetate 20 mg/0.5 mL utilizing the autoject 2 device for four weeks (Period 2).
Arm/Group | Period 1: Glatiramer Acetate 20 mg/1.0 mL | Period 2: Glatirimer Actetate
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/142
Other Adverse Events (participants affected / at risk) | 0/148 | 11/142
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Glatiramer Acetate 20 mg/1.0 mL (N=148) | Period 2: Glatirimer Actetate (N=142)
Injection site reaction (General disorders) | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data